CLINICAL TRIAL: NCT06626841
Title: A Functional Fitness Training Workout Significantly Affects Pelvic Floor Strength and Muscle Activation in Female Nulliparous Athletes
Brief Title: Assessment of Pelvic Floor Strength Variables in Female Nulliparous Athletes
Acronym: FFT-PFM
Status: Completed | Type: Observational
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Celia Rodríguez Longobardo, Principal Investigator, Universidad Politecnica de Madrid
Other Study IDs: 20221125; 20221125 (Other: Universidad Politécnica de Madrid)
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Pelvic Floor Muscle Weakness; Strength; Muscle Tone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Female athletes: Female functional fitness training athletes. The participants had to be nulliparous, had been practicing FFT or weightlifting for at least 2 years, trained a minimum of 3 days/week that did not include pelvic floor exercises, and had no medical contraindications or previous pelvic floor surgeries
  Interventions: Diagnostic Test: Pelvic floor muscles contractile capacity and activation

INTERVENTIONS:
Diagnostic Test: Pelvic floor muscles contractile capacity and activation — An initial assessment of the pelvic floor is carried out when athletes arrive at the facility. Participants then complete a FFT workout, which consists of performing as many rounds as possible (AMRAP type) of 20 wallballs, 15 box jumps, and 10 burpees within 15 minutes. These plyometrics and load lifting exercises are chosen to fatigue the PFM and are simple to execute. The pelvic floor assessment is performed again at 3 minutes following the FFT workout.
  Measurements of the pelvic floor parameters are conducted by a specialist physiotherapist. The muscle activation and strength of the PFM are obtained using a vaginal dynamometer (i.e. pelvimeter probe fixed at a vertex with two arms that can be separated by up to 25°), connected to the Phenix USB2, Vivaltis (Pelvimètre Phenix, Vivaltis).
  Other Names: pelvic floor muscles force production; pelvic floor strength; pelvic floor muscles activation

SUMMARY:
Functional Fitness Training (FFT) is a modality that seeks to improve physical fitness and performance within several functional tasks by conducting a variety of training activities such as aerobic and metabolic conditioning, resistance training, and high impact exercises. Although there are many benefits of FFT for improving fitness and body composition, their effects on the pelvic floor are not clear, as high-impact exercises performed in FFT have been shown to cause an increase in intra-abdominal pressure. When these exercises are performed repeatedly, fatigue can occur within the pelvic floor muscles (PFM), which can increase the risk of developing pelvic floor dysfunctions. However, currently little is known about how FFT activities acutely affect the PFM and whether such training regimes may contribute to long-term urinary incontinence in female FFT athletes. Therefore, this study aimed to analyse the acute effects of a FFT.workout on pelvic floor strength and muscle activation in nulliparous female FFT athletes. It is hypothesized that both strength and PFM activation of the female athletes would be reduced after a FFT workout due to PFM fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Have been practicing FFT or weightlifting for at least 2 years
* Train a minimum of 3 days/week that did not include pelvic floor exercises
* Have no medical contraindications or previous pelvic floor surgeries

Exclusion Criteria:

* Any criterion that fails to meet the inclusion criteria

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Madrid, members of a FFT facility.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Muscle activation | Change from baseline to the end of the workout, around 1 hour.
  To assess muscle activation, a vaginal dynamometer (pelvimeter probe fixed at a vertex with two arms that can be separated by up to 25°), connected to the Phenix USB2, Vivaltis (Pelvimètre Phenix, Vivaltis) is used. For the pelvic floor examination the physiotherapist introduces the closed pelvimeter inside the vagina with the supporting arm against the posterior face of the symphysis pubis. Once introduced, the probe is opened by 5º and the basal muscle activation (initial inertia index) and shock absorption (the capacity of the pelvic floor to withstand stress) are recorded.
Strength | Change from baseline to the end of the workout, around 1 hour.
  Maximal, minimum and medium force production of the pelvic floor muscles. The physiotherapist introduces the closed pelvimeter inside the vagina with the supporting arm against the posterior face of the symphysis pubis. Once introduced, the physiotherapist fixed the arms of the probe at 5º with the athlete performing a pelvic floor contraction for 10 seconds against the arms (isometric contraction). A follow-up 10-second contraction is performed after a 20-second rest to assess PFM submaximal force.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be used in anonymous form.